CLINICAL TRIAL: NCT01890538
Title: Comparison of Efficacy Between Piracetam and Dimenhydrinate in Patients With Peripheral Vertigo: A Double Blind Randomized Clinical Trial
Brief Title: Comparison of Efficacy Between Piracetam and Dimenhydrinate in Patients With Peripheral Vertigo
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Nurettin Özgür Doğan, Assistant Professor, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KOU KAEK 2013/174
Record Dates: First submitted 2013-06-25; First posted 2013-07-01 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2014-05

CONDITIONS: Peripheral Vertigo
Keywords: vertigo; dimenhydrinate; piracetam
MeSH Terms: conditions — Vertigo

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Piracetam (Active Comparator): 2 g intravenous piracetam
  Interventions: Drug: 2 g piracetam intravenous
- Dimenhydrinate (Active Comparator): Dimenhydrinate 100 mg intravenous
  Interventions: Drug: Administration of 100 mg dimenhydrinate intravenous

INTERVENTIONS:
Drug: Administration of 100 mg dimenhydrinate intravenous
  Arms: Dimenhydrinate
Drug: 2 g piracetam intravenous
  Arms: Piracetam

SUMMARY:
This study aims to investigate efficacy of two different intravenous drugs (dimenhydrinate and piracetam) in the symptomatic management of peripheral vertigo.

The patients will be randomized in two groups according to symptomatic treatment modalities: Dimenhydrinate (100 mg) and piracetam (2 g) will be given in 100 cc normal saline in 30 minutes. Each patient will be asked if her/his vertigo symptoms resolved or not, according to a numeric rating scale (0=no vertigo, 10=worst possible vertigo). The patient will be rate the intensity of symptoms in the following times:

* Numeric rating scale (1 to 10): Admission
* Numeric rating scale (1 to 10): After the study drug (No ambulation)*
* Numeric rating scale (1 to 10): After the study drug (Ambulation)*

  * Ambulation refers to head movements or walking in the room, if applicable.

ELIGIBILITY:
Inclusion Criteria:

* Presenting to emergency department with vertigo symptoms
* Adult patients (over 18)
* Agree to participate to study (understanding the study protocol and signing the informed consent form)

Exclusion Criteria:

* Patients under 18 years
* Patients diagnosed with ischemic/hemorrhagic stroke after neuroimaging
* Patient diagnosed with transient ischemic attack
* Pregnants
* Patients taking any analgesics or antihistaminic drugs last 24 hours
* Documented or declared allergy to dimenhydrinate, piracetam or benzodiazepines
* Patients who do not agree to participate to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2013-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change in numeric rating scale | Change from baseline in numeric rating scale at 30th minute

CONTACTS AND LOCATIONS:
Overall Officials: Nurettin Özgür Doğan, M.D., Assistant Professor, Principal Investigator — Kocaeli University
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)

REFERENCES:
- [Background] Scholtz AW, Schwarz M, Baumann W, Kleinfeldt D, Scholtz HJ. Treatment of vertigo due to acute unilateral vestibular loss with a fixed combination of cinnarizine and dimenhydrinate: a double-blind, randomized, parallel-group clinical study. Clin Ther. 2004 Jun;26(6):866-77. doi: 10.1016/s0149-2918(04)90130-0. PMID 15262457
- [Derived] Dogan NO, Avcu N, Yaka E, Yilmaz S, Pekdemir M. Comparison of the therapeutic efficacy of intravenous dimenhydrinate and intravenous piracetam in patients with vertigo: a randomised clinical trial. Emerg Med J. 2015 Jul;32(7):520-4. doi: 10.1136/emermed-2014-204006. Epub 2014 Jul 22. PMID 25052217
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/?term=11020677